CLINICAL TRIAL: NCT05919199
Title: The Efficiency of 18F-FDG PET Probe Signal in Bone Marrow for Predicting Acute Myeloid Leukemia Patients' Response to Induction Therapy
Brief Title: PET Tracer Based FDG Signal for Predicting Prognosis in Acute Myeloid Leukemia
Acronym: FDG-PETAML
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Hui Zeng, Director of Hematology Department of the First Affiliated Hospital of Jinan University, First Affiliated Hospital of Jinan University
Other Study IDs: MR-44-23-012821
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Bone marrow micro-environment; 18F-fluorodeoxyglucose; cancer metabolism
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AML patients, de novo or refractory/relapsed: The investigators will collect bone marrow cells under standard clinical work-up after 18F-FDG PET/CT scan and correlate the FDG signal with extramedullary infiltration, histopathological, genomics features of the patients to explore the prognostic value of FDG signal in AML.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to evaluate the predictive value of 18F-FDG PET probe signal in de novo diagnosed or refractory/relapsed patients with acute myeloid leukemia. It is hypothesized that the intensity of 18F-FDG signal, an indicator of glucose uptake capacity, in various cell subsets of bone marrow will improve the predictive effect of clinical standard prognostic work-up.

DETAILED DESCRIPTION:
Rationale:

FDG is incorporated by leukemia cells and other cell subsets in bone marrow micro-environment of various degree. The heterogeneous FDG uptake is a promising marker for predicting response to treatment. The investigators will collect bone marrow under standard clinical work-up after 18F-FDG PET/CT scan and correlate the FDG signal intensity with clinical and genomics features of the patients to explore its prognostic significance.

Objective:

The primary objective of this research project is to investigate the intensity of FDG PET probe based glucose uptake signal in predicting induction treatment response of AML. As secondary objectives, this analysis will be applied to calculate the overall predictive specificity and sensitivity of FDG probe avidity in predicting PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute myeloid leukemia, non APL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients voluntarily participated in this study and signed the informed consent

Exclusion Criteria:

* Pregnant
* Uncontrolled systemic diseases (such as diabetes, non controlled heart failure, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AML patients in First Affiliated Hospital of Jinan University
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission rate (CRc) | At the end of Cycle 2 (each cycle is about 28 days)
  Partial response (PR) + complete response (CR) rate

SECONDARY OUTCOMES:
Progress-free survival (PFS ) | From date of diagnosis until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Relapse or death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zeng, Study Chair — First Affiliated Hopital of Jinan University
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No